CLINICAL TRIAL: NCT01951911
Title: Low-dose Ketamine as Adjuvant Treatment to Morphine in Neuropathic Cancer Pain
Brief Title: Effectiveness of Ketamine in Malignant Neuropathic Pain Relief
Acronym: KETA-1
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor patient recruitment. Vast majority of the patients have exclusions criteria
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012/539
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Pain, Intractable
Keywords: Pain Management; Ketamine; Palliative care
MeSH Terms: conditions — Pain, Intractable; Agnosia | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Active Comparator): Ketamine 1 mg per kg per 24 hours as subcutaneous infusion via syringe driver for 48 hours.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Sodium chloride 0.9% administered as a subcutaneous infusion via syringe driver for 48 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Patients will receive either ketamine as subcutaneous infusion or placebo as subcutaneous infusion. The results will be compared with each other.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Placebo
  Other Names: Sodium chloride 0.9%
  Arms: Placebo

SUMMARY:
To see whether the addition of low-dose ketamine to a subcutaneous morphine infusion improves analgesia in patients with neuropathic cancer pain.

DETAILED DESCRIPTION:
Patients with cancer pain judged to have a neuropathic component and receiving pain treatment with a subcutaneous infusion of morphine will be included in a randomized, double blind, placebo-controlled, crossover study. All patients will be recruited from hospital wards (Haukeland University Hospital, Bergen). In the case of patient withdrawal or dropout, new patients will be recruited so that the total number of patients completing the study will be 20. Data from patients not completing the study will solely be used to provide information about adverse effects.

The basic treatment with subcutaneous morphine infusion will be supplemented with a separate subcutaneous infusion of ketamine 1 mg/kg/ 24 hours or NaCl 9 mg/ml (placebo).

After 48 hours (phase 1) there will be a "wash-out" period of minimum 10 hours to minimize carryover effects before the treatment is replaced by the alternative treatment for a further 48 hours (phase 2) in a standard crossover design. The treatment duration is based on ketamine's short plasma half-life which is less than 2 hours after initial equilibration.

Pain intensity (using NRS) will be recorded at rest and on movement x 4 daily. Rescue medication in the form of morphine subcutaneous bolus may be given to the patient as required. There will be a" lockout" time of 1 hour which means that the rescue dose of morphine can be repeated every 60 minutes if necessary, providing the patient is awake and has a respiratory rate of 8 or more per minute.Randomization will be performed by Haukeland University Hospital Pharmacy. The study drug/ placebo will also be prepared by the hospital pharmacy according to a standard instruction.

ELIGIBILITY:
Inclusion Criteria:

Age 18-70 years. In-patient. Cancer pain judged to have a neuropathic component. Clinically normal renal and hepatic function. Able to cooperate and understand information. Worst pain at rest or on movement 5 or more (NRS 0-10). Pain currently treated with continuous subcutaneous morphine infusion. The daily morphine dose is 48mg or more per 24 hours and a 30% increase in the daily dose has not provided sufficient pain relief.

Not treated with ketamine during the last 48 hours prior to inclusion.

-

Exclusion Criteria:

Reduced renal or hepatic function. Suspicion of morphine toxicity (sedation, hallucination, myoclonus, increasing pain).

Increased intracranial pressure (suspicion of cerebral metastases) or cerebral metastases.

Unable to cooperate/ understand information. Worst pain at rest or on movement less than 5 on NRS. Current treatment with other opioids than morphine. The patient is undergoing radiotherapy in the pain area, or has received radiotherapy in the pain area within the last four weeks.

Changes in the use of analgesics (paracetamol, NSAIDS), adjuvant drugs (antidepressants, antiepileptic, corticosteroids, muscle relaxants) or their dosages less than 2 days prior to inclusion or during the study period.

Pregnant and lactating women. Any situation in which an increase in blood pressure would constitute a hazard. Acute intermittent porphyria. Psychiatric illness, epilepsy, alcoholism, glaucoma. Hypersensitivity to any of the drugs ingredients. Current treatment with ketamine.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity compared to baseline. | 5 days
  Significant reduction in cancer pain intensity will be defined as at least 30% reduction in Numeric Rating Scale (NRS) score compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Rae F Bell, M.D. PhD., Principal Investigator — Pain Clinic, Haukeland University Hospital, 5021 Bergen, Norway
Locations (1):
- Haukeland University Hospital, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mao J, Price DD, Mayer DJ. Mechanisms of hyperalgesia and morphine tolerance: a current view of their possible interactions. Pain. 1995 Sep;62(3):259-274. doi: 10.1016/0304-3959(95)00073-2. PMID 8657426
- [Background] Ko SW, Wu LJ, Shum F, Quan J, Zhuo M. Cingulate NMDA NR2B receptors contribute to morphine-induced analgesic tolerance. Mol Brain. 2008 Jun 17;1:2. doi: 10.1186/1756-6606-1-2. PMID 18803856
- [Background] Mayer DJ, Mao J, Price DD. The association of neuropathic pain, morphine tolerance and dependence, and the translocation of protein kinase C. NIDA Res Monogr. 1995;147:269-98. PMID 8742791
- [Background] Qi X, Evans AM, Wang J, Miners JO, Upton RN, Milne RW. Inhibition of morphine metabolism by ketamine. Drug Metab Dispos. 2010 May;38(5):728-31. doi: 10.1124/dmd.109.030957. Epub 2010 Feb 2. PMID 20124399
- [Background] Bell RF, Eccleston C, Kalso E. Ketamine as adjuvant to opioids for cancer pain. A qualitative systematic review. J Pain Symptom Manage. 2003 Sep;26(3):867-75. doi: 10.1016/s0885-3924(03)00311-7. PMID 12967737
- [Background] Bell RF. Low-dose subcutaneous ketamine infusion and morphine tolerance. Pain. 1999 Oct;83(1):101-3. doi: 10.1016/s0304-3959(99)00096-2. PMID 10506678
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849
- [Background] Hagelberg NM, Peltoniemi MA, Saari TI, Kurkinen KJ, Laine K, Neuvonen PJ, Olkkola KT. Clarithromycin, a potent inhibitor of CYP3A, greatly increases exposure to oral S-ketamine. Eur J Pain. 2010 Jul;14(6):625-9. doi: 10.1016/j.ejpain.2009.10.003. Epub 2009 Nov 7. PMID 19897389
- [Background] Nisbet AT, Mooney-Cotter F. Comparison of selected sedation scales for reporting opioid-induced sedation assessment. Pain Manag Nurs. 2009 Sep;10(3):154-64. doi: 10.1016/j.pmn.2009.03.001. PMID 19706353
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771